CLINICAL TRIAL: NCT06674291
Title: Registry on the Effectiveness and Safety of the 9-month MDR-END Treatment Regimen (Delamanid, Linezolid, Levofloxacin, Pyrazinamide) in Korean Patients with Fluoroquinolone-Sensitive Pulmonary Multi-Drug Resistant Tuberculosis (MDR-TB) : a Non-interventional, Prospective Observational Study (MDR-END Registry)
Brief Title: Registry on the Effectiveness and Safety of the 9-month MDR-END Treatment Regimen in Korean Patients with FQ-sensitive MDR-TB (MDR-END Registry)
Status: Not yet recruiting | Type: Observational
Sponsor: Korea Otsuka Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: 242-402-00031
Record Dates: First submitted 2024-11-03; First posted 2024-11-05 (Actual); Last update posted 2024-11-05 (Actual); Status verified 2024-10

CONDITIONS: Tuberculosis, Multidrug-Resistant
MeSH Terms: conditions — Tuberculosis, Multidrug-Resistant | interventions — Observation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- MDR-END regimen treatment group: 1. Treatment Regimen
     Delamanid 100 mg twice daily Linezolid 600 mg once daily for the first 2 months, 300 mg once daily afterward Levofloxacin (body weight ≤ 50 kg) 750 mg once daily (body weight > 50 kg) 1000 mg once daily Pyrazinamide (body weight < 50 kg) 1000 mg once daily (body weight 50 to 70 kg) 1500 mg once daily (body weight > 70 kg) 2000 mg once daily
  2. Treatment period : 9 month (40 weeks) If the sputum test results show conversion within 3-6 months after the start of treatment, the overall treatment period is extended by 3 months for a total of 12 months (52 weeks).
  Interventions: Drug: No intervention (observational study)

INTERVENTIONS:
Drug: No intervention (observational study) — This is an observational registry conducted in the real world clinical setting and there is no intervention in this study. Treatment of MDR-END Regimen and the follow-up of subjects will be conducted in the clinical judgment of the investigator.

SUMMARY:
This study is to evaluate the effectiveness and safety of a 9-month MDR-END regimen as a treatment for fluoroquinolone-sensitive multidrug resistant pulmonary tuberculosis in the real-world clinical setting.

It will be conducted as a non-interventional, prospective, single group, multicenter design.

Subjects who are considered to meet the inclusion /exclusion criteria will receive MDR-END regimen for 9 months (or 12 months) during the treatment period according to the 5th edition of the Korean Guidelines for Tuberculosis, and will be followed-up for 12 months after the end of treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Adults aged 19 years or older who have been diagnosed with multidrug resistant pulmonary tuberculosis
2. Adults prescribed MDR-END regimen according to the Korean Guidelines for Tuberculosis after being informed of this study from the investigator and signing an informed consent form

Exclusion Criteria:

1. Patients with confirmed quinolone resistance
2. Patients with hypersensitivity to one or more of the following drugs: Delamanid, Linezolid, Levofloxacin, and Pyrazinamide
3. Patients who are found to have contraindications according to the approved labels of Delamanid, Linezolid, Levofloxacin, or Pyrazinamide
4. Patients with or with a history of optic neuritis or peripheral neuritis
5. Patients with genetic problems such as galactose intolerance, Lapp lactase deficiency, or glucose-galactose malabsorption
6. Pregnant or lactating women
7. Women of childbearing potential who are unwilling to use appropriate contraception during the study treatment

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 222 adult men and women with fluoroquinolone-sensitive multidrug resistant pulmonary tuberculosis will be enrolled in this study.
  To determine the sample size of this study, the treatment success rate of the study group in the MDR-END trial treated with Delamanid, Linezolid, Levofloxacin, and Pyrazinamide to shorten the treatment duration of multidrug resistant tuberculosis in patients with fluoroquinolone-sensitive multidrug resistant tuberculosis was assumed to be the expected effectiveness rate.
  The treatment success rate of the study group in the MDR-END trial was 84.72% according to the 5th edition of the Korean Guidelines for Tuberculosis, and the number of subjects required was 222 subjects calculated with a 95% confidence interval, 5% tolerance and 10% dropout rate.
Sampling Method: Non-Probability Sample
Enrollment: 222 (Estimated)
Dates: Start 2024-11-30 (Estimated); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Treatment success rate at the end of treatment | At the end of treatment
  "Cured" and "Treatment Completed" from the result of multidrug resistant pulmonary tuberculosis treatment are defined as treatment success, and the treatment outcomes of multidrug resistant pulmonary tuberculosis treatment are determined according to the 5th edition of the Korean Guidelines for Tuberculosis.

SECONDARY OUTCOMES:
Treatment success rate at 12 months after the end of treatment (end of study) | At 12 months after the end of treatment (end of study)
Recurrence rate after treatment success | During follow up period (12 months after the end of treatment)
Treatment-emergent adverse events (TEAEs) | During the treatment period and up to one month after the end of treatment
TEAEs by severity | During the treatment period and up to one month after the end of treatment
Mortality and time to death | During the treatment period and up to one month after the end of treatment
TEAEs related to QT prolongation | During the treatment period and up to one month after the end of treatment

IPD SHARING:
Plan to Share IPD: No